CLINICAL TRIAL: NCT01408134
Title: Viability Imaging in Volumetric Angiography (VIVA 1): A Single Center Trial of the Detection of Delayed Hyperenhancement on CT Angiography
Brief Title: Viability Imaging in Volumetric Angiography (VIVA 1)
Acronym: VIVA 1
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI/Project director no longer at facility
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VIVA 1
Record Dates: First submitted 2011-07-28; First posted 2011-08-03 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Myocardial Scarring
Keywords: Inter-reader variability of myocardial viability imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: DE CT — Delayed scan (per VIVA protocol): The delayed scan will be performed 10 minutes after contrast second contrast bolus complete using axial acquisition at 100 kVp. Scan length will be limited to the cardiac structures.

SUMMARY:
The primary objective of this study is twofold:

1. To define inter-reader variability of myocardial viability imaging within the first pass and delayed enhancement cardiac CT perfusion imaging
2. To evaluate DE CT image quality using a consensus DECT protocol

DETAILED DESCRIPTION:
The presence of myocardial scar using radionuclide or magnetic resonance imaging techniques indicates myocardial segments with a reduced likelihood of functional recovery following myocardial revascularization. Preliminary evidence suggests that multi-detector CT (MDCT) angiography also can detect irreversible myocardial scarring through the detection of regions of delayed hyperenhancement (DE) of the myocardium.1-4 However, existing studies have been performed in single centers, and the reproducibility, and impact of this modality on recovery of myocardial function is unknown. In this study, the investigators propose a single-center trial using a standardized MDCT DE protocol among patients scheduled for clinical cardiac CT with planned reoperative surgical. The primary endpoint will be characteristics of DE imaging of the myocardium including its inter-reader variability and factors associated with image quality. These findings will further our understanding of the role of DE MDCT for the detection of myocardial viability.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be adults, ages 18 and above with:

  1. Known CAD with prior MI based upon clinical history or electrocardiographic criteria
  2. Planned redo-surgical myocardial revascularization
  3. Referred for CT (and eligible) for pre-op substernal mapping/coronary artery evaluation

Exclusion Criteria:

1. Inability to provide informed consent
2. Allergy to iodinated contrast media (unless pre-medicated with medical prophylaxis)
3. Chronic kidney disease manifested by a serum creatinine >1.5 mg/dL, an estimated creatinine clearance <50 ml/kg/min or on dialysis
4. Currently reporting or evaluated in NYHA class IV heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Inter-reader variability of myocardial viability | day One
  To define inter-reader variability of myocardial viability imaging within the first pass and delayed enhancement cardiac CT perfusion imaging, specifically:
  * Per myocardial segment binary visual estimation of the presence/absence of contrast enhancement on either a first pass or 10-minute delayed CT scan.
  * Myocardial enhancement (hyper and hypo-enhancement) will be evaluated using a binary assessment for estimation of the involved myocardial segments on delayed images. Regional wall motion will be assessed qualitatively using a 4 point scale: normal, hypokinetic, akinetic, dyskinetic.
DE CT image quality | day One
  To evaluate DE CT image quality using a consensus DECT protocol

SECONDARY OUTCOMES:
Scan and patient factors related to the image quality | day One
  The secondary endpoint will be to describe the scan and patient factors related to the image quality on myocardial CT perfusion imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States